CLINICAL TRIAL: NCT00186251
Title: Use of High Dose Chemotherapy Followed by Peripheral Blood Stem Cell Rescue for Relapsed or Resistant Hodgkin's Disease
Brief Title: High Dose Chemotherapy Followed By PBSC Rescue for HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT24; BMT24; NCT00186251; 13322 (Other: Stanford IRB)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-07

CONDITIONS: Hodgkin Disease
MeSH Terms: conditions — Hodgkin Disease

INTERVENTIONS:
Procedure: high dose chemo then auto hematopoietic cell transplant

SUMMARY:
To evaluate the role of high dose chemotherapy with autologous hematopoietic cell transplantation in the treatment of Hodgkin's Disease.

DETAILED DESCRIPTION:
Use of High Dose Chemotherapy Followed by Peripheral Blood Stem Cell Rescue for Relapsed or Resistant Hodgkin's Disease

ELIGIBILITY:
Inclusion Criteria:- adequate organ function

* recurrent HD Exclusion Criteria:- CNS disease
* no prior malignancy

Ages: 4 Weeks to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1998-03; Study Completion 2005-07

PRIMARY OUTCOMES:
Overall survival
FFS
Response rates

SECONDARY OUTCOMES:
Toxicity of high dose chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Sally Arai, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States